CLINICAL TRIAL: NCT00627744
Title: Phase IV Study Evaluating the Effect of Sitagliptin (Januvia™) on Beta-cell Function in Patients With Acute Myocardial Infarction or Unstable Angina Pectoris and Newly Detected Impaired Glucose Tolerance or Type 2 Diabetes.
Brief Title: Beta-cell Function in Glucose Abnormalities and Acute Myocardial Infarction
Acronym: BEGAMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars Ryden, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEGAMI
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Infarction; Unstable Angina Pectoris; Diabetes Mellitus; Impaired Glucose Tolerance
Keywords: Type 2 diabetes, IGT, Myocardial infarction, Incretins
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Diabetes Mellitus; Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BE 1 (Placebo Comparator): Patients in this arm are randomly assigned to treatment with placebo
  Interventions: Drug: Sitagliptin
- BE 2 (Active Comparator): Patients in this arm are randomly assigned to treatment with Sitagliptin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — BE 1 receives Placebo tablets od during 12 weeks BE 2 receives Sitagliptin tablets 100 mg od during 12 weeks
  Other Names: Active drug is Januvia produced by Merck

SUMMARY:
A three months, double-blind, randomised, parallel-group study evaluating the efficacy of sitagliptin (Januvia™) versus placebo on beta-cell function in patients with newly detected glucose abnormalities and acute myocardial infarction or unstable angina pectoris.

Primary endpoint Improvement in beta-cell function measured by means of the insulinogenic index (ΔI30/ΔG30) obtained from an oral glucose tolerance test (OGTT).

Secondary endpoints

1. Improvement of glucose tolerance by means of an OGTT
2. Improvement in endothelial function
3. Improvement in incretin-independent beta-cell function measured as the Acute Insulin Response (ΔAIRG) during an intravenous glucose tolerance test

DETAILED DESCRIPTION:
GENERAL AIM / PRIMARY OBJECTIVE The primary objective is to show that sitagliptin (Januvia™) 100 mg once daily for three months improves beta-cell function in patients with AMI or unstable angina pectoris and newly discovered glucose abnormalities (IGT or T2DM).

PRIMARY ENDPOINT The primary endpoint is improvement in beta-cell function after three months treatment measured by means of insulinogenic index (ΔI30/ΔG30) obtained from an oral glucose tolerance test (OGTT).

SECONDARY ENDPOINTS

1. Improvement of glucose tolerance tested with an OGTT after three months.
2. Improvement in endothelial function (measured with Endo-PAT2000, Itamar) after three months.
3. Improvement in GLP-1 independent beta-cell function after three months measured as the ΔAIRG obtained from a "Frequently sampled intravenous glucose tolerance test" (FSIGT).

NUMBER OF PATIENTS PLANNED A total of 70-80 consecutive patients will be included with 35-40 patients in each treatment arm.

TREATMENTS TO BE COMPARED Active substance: Sitagliptin Januvia™ 100 mg once daily orally during three months

Comparator drug Placebo

CONCOMITANT THERAPY All patients should receive evidence based treatment for secondary prevention of coronary heart disease according to the most recent ESC guidelines [60,61].

All patients will receive structured life style intervention strategies according to local practise.

EFFICACY The primary endpoint is improvement in beta-cell function after three months treatment measured by means of insulinogenic index (ΔI30/ΔG30) obtained from an oral glucose tolerance test (OGTT).

Secondary endpoints

1. Improvement of glucose tolerance tested with an OGTT after three months.
2. Improvement in endothelial function (measured with Endo-PAT2000, Itamar) after three months.
3. Improvement in GLP-1 independent beta-cell function after three months measured as the ΔAIRG obtained from a "Frequently sampled intravenous glucose tolerance test" (FSIGT).

Methodology OGTT: Oral administration of 75 g of Glucose in 200 ml water with lemon extract is administered on the morning following an overnight fast of 12 hours A capillary blood glucose curve is obtained during 2 hours (just before and at 30, 60, 90 and 120 minutes after the glucose ingestion).

Endo-PAT2000: The Endo-PAT2000 is a non-invasive device for non-invasive characterisation of endothelial function and dysfunction and arterial stiffness. The endothelial function assessment is based on the endothelial mediated arterial response (at the level of a distal phalanx of a finger) to a five-minute occlusion of the brachial artery.

FSIGT: The patient is investigated on the morning after an overnight fast. A catheter will be inserted into an antecubital vein for blood sampling and into a contralateral antecubital vein for glucose injection. Basal samples will be drawn at 10 and at 1 min. At time 0, glucose (300 mg/kg) will be injected during 1 min, and then additional samples will be collected at 3, 4, 5, 6, 8, 10, 15, 20, 25, 30, 40, 60, 80, 100, 120, 150, and 180 min [62].

INVESTIGATIONAL PLAN This is a three months, double-blind, randomised, parallel-group study evaluating the efficacy of sitagliptin (Januvia™) versus placebo on beta-cell function in patients with AMI or unstable angina pectoris with newly discovered glucose abnormalities (IGT + T2DM).

SAMPLE SIZE ISSUES The assumption for the sample size calculation is based on a previous study from our group where the insulinogenic index was measured in patients with AMI and newly discovered type 2 diabetes and IGT [21]. The mean and standard-deviation of the ΔAIRG are estimated to 50 ± 35 (pmol/mmol). To detect an increase of 50 % between the two treatment groups at a 5 % level of significance with 80 % power using a two-tailed t-test, a sample size of 64 patient would be necessary (PROC POWER in SAS 9.1.3). With an an additional 5 % to be able to use non-parametric methods the total sample size is set to 70 patients.

ETHICS AND REGULATORY The trial will not be initiated until the protocol and informed consent and subject information form have been reviewed and received approval from the local ethics committee.

Informed Consent and Subject Information Each patient should receive oral and written information. Patients will be included following oral and written consent. Patient data will be protected and patients will be insured by Swedish law. All patients must be informed that they, whenever they wish, may withdraw from the study and that they in case of withdrawal will be treated according to the best possible routine standards of the centre.

QUALITY ASSURANCE AUDIT Monitoring visits will be performed before inclusion of first subject, regularly during trial conduct and after data based closed in collaboration with the Karolinska Clinical Research Trial and Support Centre. The investigators will permit trial-related monitoring, audits, IRB/IEC reviews, and regulatory inspections, providing direct access to source data/documents.

ADVERSE EVENTS All adverse events, serious and non-serious, occurring during the course of the clinical trial will be collected, documented and reported to the sponsor by the investigator. An adverse event is defined as any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

The non-serious adverse events that have been observed in patients treated with sitagliptin are (>5% incidence and greater incidence than placebo):

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with an acute myocardial infarction or unstable angina pectoris according to the joint ESC and ACC recommendations [58].
2. Classification of impaired glucose tolerance (IGT) or type 2 diabetes (T2DM) by means of an oral glucose tolerance test (OGTT) according to WHO [59].
3. Patients who have signed a written informed consent consistent with ICH-GCP guidelines and local legislations prior to participation in the trial.

Exclusion criteria:

1. No informed consent.
2. <18 years old.
3. Previous known type 2 diabetes.
4. Admission plasma glucose >12 mmol/L.
5. Impaired renal function (S-creatinine ≥ 130 μmol/L or need of renal dialysis).
6. BMI>30.
7. Known Type 1 diabetes, GAD positive or C-peptide<0.30.
8. Patients with severe concomitant disease (i.e. malignancy, liver failure).
9. Patients who at discharge are planned for Coronary Artery Bypass Grafting or percutaneous coronary intervention.
10. Congestive heart failure (NYHA III-IV).
11. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception.
12. Patients who, in the opinion of the investigator, will have difficulties to comply with the protocol (examples: alcohol or drug abuse, psychiatric disorder, resident outside of the catchment area).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Improvement in beta-cell function measured by means of the insulinogenic index (ΔI30/ΔG30) obtained from an oral glucose tolerance test (OGTT) | By the end of the study as stated

SECONDARY OUTCOMES:
Improvement of glucose tolerance by means of an OGTT | As stated for the study
Improvement in endothelial function | As stated for the study
Improvement in incretin-independent beta-cell function measured as the Acute Insulin Response (ΔAIRG) during an intravenous glucose tolerance test. | As stated for the study

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rydén, Professor, Study Chair — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Karolinska University Hospital Solna, Stockholm

REFERENCES:
- [Derived] Hage C, Lundman P, Ryden L, Mellbin L. Fasting glucose, HbA1c, or oral glucose tolerance testing for the detection of glucose abnormalities in patients with acute coronary syndromes. Eur J Prev Cardiol. 2013 Aug;20(4):549-54. doi: 10.1177/2047487312444371. Epub 2012 Mar 28. PMID 22456695